CLINICAL TRIAL: NCT05415241
Title: Exploratory Study of Aerosol Inhalation of FB2001 for Post-exposure Prophylaxis of Close Contacts of COVID-19 Patients
Brief Title: Exploratory Study of Aerosol Inhalation of FB2001 for Post-exposure Prophylaxis of COVID-19 Close Contacts
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Frontier Biotechnologies Inc. (Industry); Shanghai Center for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, Jieming QU, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: FB2001-PEP-1
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Close Contact Transmission
MeSH Terms: interventions — FB2001

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FB2001Exploratory (Experimental): Stage 1 (Exploring the dose): FB2001 once daily for 5 consecutive days. If the drug is well tolerated but efficacy is inadequate, FB2001 BID for 5 consecutive days.
  Stage 2 (Sample size expansion): FB2001 once daily or twice daily for 5 consecutive days depending on the result of stage 1.
  Interventions: Drug: FB2001

INTERVENTIONS:
Drug: FB2001 — Stage 1 (Exploring the dose): Twenty participants will be enrolled for aerosol inhalation of FB2001 once daily for 5 consecutive days. If the drug is well tolerated but efficacy is inadequate, another twenty participants will be enrolled for aerosol inhalation of FB2001 BID for 5 consecutive days.
  Stage 2 (Sample size expansion): Another twenty participants will be enrolled for aerosol inhalation of FB2001 once daily or twice daily for 5 consecutive days depending on the result of stage 1.

SUMMARY:
This is a single-arm, open-label, dose ramp-up exploratory clinical trial to evaluate the efficacy, safety and tolerance of aerosol inhalation of FB2001 as post-exposure prophylaxis among close contacts of COVID-19 patients.

This study will enroll 20 to 60 close contacts of COVID-19 patients aging 18 to 65 years.

After signing the informed consent form, the qualified subjects will be given FB2001 once or twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals aged 18-65 years.
2. COVID-19 close contacts determined by epidemiological investigation (living in the same room within 72 hours before screening with individuals having positive nucleic acid amplification test for SARS-CoV-2 ).
3. Having two consecutive negative nucleic acid tests within 72 hours before enrollment.
4. Participants of childbearing age must agree to use a highly effective method of contraception.
5. Sign the informed consent form.

Exclusion Criteria:

1. Pregnant women.
2. Participants who have history of prior drug allergy or are vulnerable to allergy.
3. Participants who infected with SARS-CoV-2 within previous 6 months.
4. Fever (body temperature > 38 ℃), frequent cough and other symptoms suggestive of COVID-19 upon screening.
5. Participants with a history of asthma or chronic obstructive pulmonary disease.
6. Participants with known history of active liver disease, acute kidney disease or chronic kidney disease.
7. Participants with known history of stroke (except cavity infarction), serious heart disease or myocardial infarction.
8. Participants with known diagnosis of Alzheimer's disease, Parkinson's disease or tumor (except for radical tumor resection).
9. Blood pressure >180/100mmHg at screening.
10. Participated in other interventional studies within previous 6 months.
11. Uptaking CYP3A4/5 strong inducers or inhibitors (rifampicin, phenytoin, carbamazepine, St. John's wort, clarithromycin, itraconazole, ketoconazole, ritonavir, cobicistat, darunavir, atazanavir, lopinavir, nelmatevir, nefazodone, etc.).
12. Participants who need to use other anti-SARS-CoV-2 therapeutic drugs during the study period.
13. Other conditions are considered unsuitable to participate in the researcher after evaluation by the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-09 (Estimated); Primary Completion 2022-08-09 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
efficacy index of post-exposure prophylaxis against COVID-19 | 7 days post aerosol inhalation of FB2001
  The percentage of participants having positive nucleic acid amplification test for SARS-CoV-2 within 7 days post inhalation of FB2001.
efficacy index of post-exposure prophylaxis against COVID-19 | 14 days post aerosol inhalation of FB2001
  The percentage of participants having positive nucleic acid amplification test for SARS-CoV-2 within 14 days post inhalation of FB2001.
safety index | during aerosol inhalation of FB2001 or 30 minutes (or longer, if necessary) post aerosol inhalation of FB2001
  The number of cases of intolerance or anaphylaxis, as well as the incidence of treatment-related adverse events (TRAEs) during aerosol inhalation therapy.